CLINICAL TRIAL: NCT05163977
Title: Comparison Between Blumgart Anastomosis and Cattell Warren Anastomosis in Reduction of Post-Operative Complications After Pancreaticoduodenectomy Procedure
Brief Title: Pancreatico Enteric Anastomosis Post Pancreaticoduodenectomy
Acronym: PEAPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ehab Abdulkarim Abdulmaksoud, Assistant Lecturer of Surgical Oncology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SO2106-31005
Record Dates: First submitted 2021-07-13; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Cancer of Pancreas
Keywords: cancer pancreas; pancreatico-jejunostomy; pancreatico-enteric anasomosis; pancreatic anastomosis; post-operative pancreatic fistula; pancreaticoduodenectomy; whipple's procedure
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cattell Warren Anastomosis (Active Comparator)
  Interventions: Procedure: Cattell Warren Anastomosis
- Blumgart Anastomosis (Experimental)
  Interventions: Procedure: Blumgart Anastomosis

INTERVENTIONS:
Procedure: Blumgart Anastomosis — The anti-mesenteric border of the jejunal loop proximal to the hepatico-jejunostomy is brought against the pancreatic stump. With the pancreatic stump retracted by the stay sutures, the transected end of pancreatic duct is first identified and secured by means of a blunt tipped probe. Each trans-pancreatic, suture was performed using a single Polydioxanone (PDS) 3 -0 blunt needle. We usually take 4 sutures, 2 on each side of the duct. The process is repeated in the same manner with the remaining sutures which are tightened at the end to approximate the jejunum loop to the stump. A small stab incision is then made at the anti-mesenteric border of the jejunum and a duct to mucosa anastomosis is constructed using an interrupted 5-0 Prolene. The process is completed by placing each of the retained needles through the seromuscular layer of the anterior jejunal wall and each knot is tied over the jejunal wall which is then warped over the cut end of the stump
  Arms: Blumgart Anastomosis
Procedure: Cattell Warren Anastomosis — It is a two layer, interrupted, end to side pancreatico-jejunostomy. First an interrupted sutures between the posterior capsule and the seromuscular layer of the jejunum was constructed using PDS 3-0 , then a duct to mucosa interrupted sutures were taken using PDS 5-0 and finally interrupted sutures between the anterior capsule and the jejunum . The main difference here is that the sutures are taken in a conventional way which is tangential to the pancreatic capsule and parenchyma
  Arms: Cattell Warren Anastomosis

SUMMARY:
The aim of this study is to make a step for evaluation and presentation of a safe technique for pancreatico-jejunostomy that help in minimizing post-operative morbidity and mortality in pancreatic cancer patient by comparing Blumgart anastomosis with Cattell warren technique of anastomosis.

DETAILED DESCRIPTION:
Study Design This study is a randomized prospective clinical trial. Methods of randomization: Randomized block design

The objective of the study was to evaluate the effect of Blumgart anastomosis versus Cattell Warren techniques for pancreatico-jejunostomy regarding

* Surgical technique
* Peri-operative outcome including

  1. Length of hospital stay
  2. Post-operative pancreatic fistula
  3. ICU admission and stay
  4. Operative time
  5. Other morbidity and mortality

Data collection:

All data will be collected for each group and will be divided into Patients' factors, intraoperative and postoperative factors. Patients' factors include patients' demographics, co-morbidities, neoadjuvant treatment, Pathology and Biliary drainage. Intra-operative factors include type of Pancreaticoduodenectomy (PD) (Whether classic or PPPD), Operative time in hours and estimated blood loss in ml, pancreatic duct and texture of pancreas. Post-operative factors include the short term post-operative course which will be divided into specific complications (pancreatic leakage, biliary leakage, delayed gastric emptying, 2ry hemorrhage, intra-abdominal collection, deep wound infection, Portal Vein (PV) - Superior Mesenteric Vein (SMV) thrombosis and general surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Known Pancreatic head cancer diagnosed radiologically.
* Operable and borderline pancreatic cancer.
* Patients who will undergo upfront surgery and those who received neoadjuvant chemotherapy are included.

Exclusion Criteria:

* Metastatic patients.
* Locally advanced cases.
* Patients with comorbidities who are unfit for major surgical procedures.
* Patients with very small pancreatic duct where the pancreatic duct can't be identified.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-06-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Post-Operative Pancreatic Fistula | Up to 10 days after the operation
  We used the International Study Group of Pancreatic Fistula (ISGPF) definition which is any measurable pancreatic fluid output after postoperative day 3 (containing more than three times the normal serum amylase level; more than 300 IU/L) with clinical signs of an infection and/or necessitating a change in clinical management.

SECONDARY OUTCOMES:
Biliary leakage | Up to 10 days after the operation
  Any biliary output via percutaneous drains after the first postoperative day, or detected at a re-laparotomy
Post-Operative bleeding | 1-3 weeks
  including early and late bleeding (1-3 weeks post-operative) According to ISGPF it is defined as any bleeding from the surgical site with a drop in hemoglobin concentration greater than 3 g/dL with peripheral circulatory impairment requiring medical, surgical, or radiological intervention.
Hospital Stay | Immediate after surgery and until the discharge of the patient ,including the readmission within the first 30 days after the operation
  the post operative hospital stay
Operative Time | During the operation
  Time of the surgical procedure in hours
primary or reactionary hemorrhage | During the operation and within the first 24 hours after the operation
  Bleeding that occurs during or in the first day after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ehab A Abdulmaksoud, master, Principal Investigator — National Cancer Institute Cairo University
Locations (1):
- The Egyptian National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No